CLINICAL TRIAL: NCT02713581
Title: IgG Dependent Monocyte Activation in Proximal Venous Thromboembolism
Acronym: ActiMon
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2015/SB-01; 2016-A00447-44 (Other: RCB number)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Venous Thromboembolism; Pulmonary Embolism
Keywords: Proximal venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with proximal VTE: Patients will correspond to cases of proximal venous thromboembolism. They will be recruited during consultations conducted for the chronic management of a history of proximal venous thromboembolism or thrombophilia following a recent history of proximal venous thromboembolism. Venous thromboembolism, outside of acute phase episodes, has good symptom stability over time; no difference is to be expected between patients with a chronic history of proximal venous thromboembolism and new patients coming in for a checkup. Note that these patients may or may not have a history of placental vascular disease.
  Intervention: Blood sampling
  Interventions: Biological: Blood sampling
- Women with >1 healthy pregnancy: This populations is composed of healthy, female, adult volunteers (<50 years in age) that have had at least 1 healthy pregnancy.
  Intervention: Blood sampling
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Venous blood will be sampled for laboratory analyses (see outcomes).

SUMMARY:
The primary objective of this study is to search for, in vitro, elements associated with IgG-dependent monocyte activation (signaling pathway activation, expression of pro-coagulant and pro-inflammatory factors) and to describe their prevalence in female patients with a history of proximal venous thromboembolism (proximal deep vein thrombosis or pulmonary embolism) compared to control women.

DETAILED DESCRIPTION:
The secondary objectives of this study include to compare the IgG-dependent monocyte activation profiles as a function of laboratory thrombophilia parameters. Essentially: Is IgG-dependent cell activation associated with the presence of anti-phospholipid antibodies (or their subtypes?), or do these profiles indicate something beyond the nosology of anti-phospholipid syndrome?

ELIGIBILITY:
Inclusion Criteria for patients:

* The patient has given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Adult woman 18 to 50 years old
* At least one prior incident of proximal venous thromboembolism (proximal deep vein thrombosis or pulmonary embolism) over three months ago regardless of the patient's history of placental vascular disease

Exclusion Criteria for patients:

* The patient is participating in another interventional study, or has participated in another interventional study within the past 3 months
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or is an adult under guardianship
* It is impossible to correctly inform the patient, or the patient refuses to sign the consent
* Postmenopausal women
* Pregnancy within the last 3 months
* Isolated history of superficial venous thrombosis
* Isolated history of distal venous thrombosis
* History of malignancy (solid or hematological)
* Known positive serology for hepatitis B
* Known positive serology for hepatitis C
* Known positive serology for human immunodeficiency virus (HIV)
* Episode of inflammatory or infectious disease dating back less than 3 months
* Impaired liver function characterized by liver enzymes (Alanine aminotransferase/ Aspartate aminotransferase) greater than 3 times normal
* Impaired renal function tests characterized by a glomerular filtration rate below 80 ml / min
* Drug background therapy (other than antiplatelet or anticoagulant therapy) used in the treatment of autoimmune disease

Inclusion Criteria for healthy volunteers:

* The healthy volunteer has given her informed and signed consent
* The healthy volunteer must be insured or beneficiary of a health insurance plan
* Adult woman 18 to 50 years old
* A history of at least one normal pregnancy defined by the birth of a child born alive in the absence of placental vascular complications

Exclusion Criteria for healthy volunteers:

* The healthy volunteer is participating in another interventional study, or has participated in another interventional study within the past 3 months
* The healthy volunteer is in an exclusion period determined by a previous study
* The healthy volunteer is under judicial protection, or is an adult under guardianship
* It is impossible to correctly inform the healthy volunteer, or the healthy volunteer refuses to sign the consent
* Postmenopausal women
* Pregnancy within the last 3 months
* History of superficial venous thrombosis
* History of distal venous thrombosis
* History of malignancy (solid or hematological)
* Known positive serology for hepatitis B
* Known positive serology for hepatitis C
* Known positive serology for human immunodeficiency virus (HIV)
* Episode of inflammatory or infectious disease dating back less than 3 months
* Impaired liver function characterized by liver enzymes (Alanine aminotransferase/ Aspartate aminotransferase) greater than 3 times normal
* Impaired renal function tests characterized by a glomerular filtration rate below 80 ml / min
* Background drug treatment
* History of proximal venous thromboembolism
* History of placental vascular disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient population description: Patients will correspond to cases of proximal venous thromboembolism. They will be recruited during consultations conducted for the chronic management of a history of proximal venous thromboembolism or thrombophilia following a recent history of proximal venous thromboembolism. Venous thromboembolism, outside of acute phase episodes, has good symptom stability over time; no difference is to be expected between patients with a chronic history of proximal venous thromboembolism and new patients coming in for a checkup. Note that these patients may or may not have a history of placental vascular disease.
  Healthy volunteer population description: This populations is composed of healthy, female, adult volunteers (<50 years in age) that have had at least 1 healthy pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
The presence/absence of an activation profile | Day (0)
  The following will be taken into account: Six signaling pathways (Protein kinase B, extracellular-signal-regulated kinases, Signal transducer and activator of transcription 5, P38 mitogen-activated protein kinases, Mechanistic Target Of Rapamycin, nuclear factor kappa-light-chain-enhancer of activated B cells), increases in the expression of tissue factor, and 5 pro-inflammatory factors (Intercellular Adhesion Molecule, tumor necrosis factor alpha, interferon gamma, Interleukin-1 beta, Interleukin 8). A pathway will be considered as "activated" or an expression profile as "increased" when the observed value is superior to the 95% confidence interval determined using healthy volunteer values. A patient is considered as having an activation profile if at least one of the above pathways or expressions is considered as activated / increased.

SECONDARY OUTCOMES:
History of proximal deep vein thrombosis? yes/no | Day (0)
History of pulmonary embolism? yes/no | Day (0)
History of placental vascular pathology? yes/no | Day (0)
The presence / absence of antiphospholipid antibodies: lupus anticoagulant antibodies | Day (0)
The presence / absence of antiphospholipid antibodies: anti-cardiolipid antibodies | Day (0)
The presence / absence of antiphospholipid antibodies: anti-beta2-glycoprotein 1 antibodies | Day (0)
The presence / absence of a constitutional biological thrombophilia | Day (0)
  The presence / absence of a constitutional biological thrombophilia (mutation of the Leiden V factor and the prothrombin gene, deficiency in physiological coagulation inhibitors)
Fibrin monomer (blood; mg/ L) | Day (0)
Blood D-dimers (ng/mL) | Day (0)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Bouvier, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes